CLINICAL TRIAL: NCT00809848
Title: Safety and Efficacy of AGN 210669 Ophthalmic Solution in Patients With Ocular Hypertension or Primary Open-Angle Glaucoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 210669-003
Record Dates: First submitted 2008-12-16; First posted 2008-12-17 (Estimated); Results first posted 2013-10-18 (Estimated); Last update posted 2013-10-18 (Estimated); Status verified 2013-08

CONDITIONS: Ocular Hypertension; Glaucoma
MeSH Terms: conditions — Ocular Hypertension; Glaucoma | interventions — Bimatoprost

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- AGN-210669 ophthalmic solution, 0.075% (Experimental): AGN-210669 non-preserved ophthalmic solution, 0.075%. One drop in both eyes each morning once-daily for 2 weeks.
  Interventions: Drug: AGN-210669 ophthalmic solution, 0.075%
- AGN-210669 ophthalmic solution, 0.05% (Experimental): AGN-210669 non-preserved ophthalmic solution, 0.05%. One drop in both eyes each morning once-daily for 2 weeks.
  Interventions: Drug: AGN-210669 ophthalmic solution, 0.05%
- AGN-210669 ophthalmic solution, 0.025% (Experimental): AGN-210669 non-preserved ophthalmic solution, 0.025%. One drop in both eyes each morning once-daily for 2 weeks.
  Interventions: Drug: AGN-210669 ophthalmic solution, 0.025%
- bimatoprost ophthalmic solution 0.03% (Active Comparator): Bimatoprost ophthalmic solution 0.03%. One drop in both eyes each morning once-daily for 2 weeks.
  Interventions: Drug: bimatoprost ophthalmic solution 0.03%
- AGN-210669 vehicle ophthalmic solution (Placebo Comparator): AGN-210669 vehicle non-preserved ophthalmic solution. One drop in both eyes each morning once-daily for 2 weeks.
  Interventions: Drug: AGN-210669 vehicle ophthalmic solution

INTERVENTIONS:
Drug: AGN-210669 ophthalmic solution, 0.075% — AGN-210669 non-preserved ophthalmic solution, 0.075%. One drop in both eyes each morning once-daily for 2 weeks.
  Arms: AGN-210669 ophthalmic solution, 0.075%
Drug: AGN-210669 ophthalmic solution, 0.05% — AGN-210669 non-preserved ophthalmic solution, 0.05%. One drop in both eyes each morning once-daily for 2 weeks.
  Arms: AGN-210669 ophthalmic solution, 0.05%
Drug: AGN-210669 ophthalmic solution, 0.025% — AGN-210669 non-preserved ophthalmic solution, 0.025%. One drop in both eyes each morning once-daily for 2 weeks.
  Arms: AGN-210669 ophthalmic solution, 0.025%
Drug: bimatoprost ophthalmic solution 0.03% — Bimatoprost ophthalmic solution 0.03%. One drop in both eyes each morning once-daily for 2 weeks.
  Other Names: Lumigan®
  Arms: bimatoprost ophthalmic solution 0.03%
Drug: AGN-210669 vehicle ophthalmic solution — AGN-210669 vehicle non-preserved ophthalmic solution. One drop in both eyes each morning once-daily for 2 weeks.
  Arms: AGN-210669 vehicle ophthalmic solution

SUMMARY:
The study will evaluate the safety and efficacy of AGN-210669 ophthalmic solution in comparison with AGN-210669 vehicle and bimatoprost ophthalmic solution dosed once-daily each morning, in subjects with ocular hypertension or primary open-angle glaucoma. Subjects will be followed for 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Ocular hypertension or primary open-angle glaucoma
* Females of non-childbearing potential
* Subject requires IOP-lowering therapy in both eyes
* IOP ≥ 22 mm Hg and ≤ 34 mm Hg
* Has a visual acuity score of 20/100 or better in each eye

Exclusion Criteria:

* Uncontrolled systemic disease
* Active ocular disease
* Alteration of existing chronic systemic medications
* Known allergy or sensitivity to the study medications
* Ophthalmic corticosteroids
* Visual field loss which in the opinion of the investigator is functionally significant
* History of ocular laser, intraocular surgery, or refractive surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2009-02; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Artesia, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AGN-210669 Ophthalmic Solution, 0.075% | AGN-210669 Ophthalmic Solution, 0.05% | AGN-210669 Ophthalmic Solution, 0.025% | Bimatoprost Ophthalmic Solution 0.03% | AGN-210669 Vehicle Ophthalmic Solution
Started | 36 | 34 | 34 | 31 | 37
Completed | 36 | 34 | 34 | 30 | 34
Not Completed | 0 | 0 | 0 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AGN-210669 Ophthalmic Solution, 0.075% | AGN-210669 Ophthalmic Solution, 0.05% | AGN-210669 Ophthalmic Solution, 0.025% | Bimatoprost Ophthalmic Solution 0.03% | AGN-210669 Vehicle Ophthalmic Solution | Total
Number analyzed (Participants) | 36 | 34 | 34 | 31 | 37 | 172
Age, Customized [Number; unit: Participants]
  <45 years | 1 | 0 | 2 | 1 | 3 | 7
  Between 45 and 65 years | 23 | 20 | 18 | 18 | 18 | 97
  >65 years | 12 | 14 | 14 | 12 | 16 | 68
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 18 | 21 | 20 | 20 | 101
  Male | 14 | 16 | 13 | 11 | 17 | 71

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average Eye Intraocular Pressure (IOP)
Description: IOP is a measurement of the fluid pressure inside the eye. The average of the 2 eyes is used for the analyses. A negative number change from baseline indicates a reduction in IOP (improvement) and a positive number change from baseline indicates an increase in IOP (worsening).
Time Frame: Baseline, Day 14 Hour 0
Population: Modified Intent to Treat: all randomized and treated patients who had at least a baseline visit and 1 postbaseline IOP evaluation
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury (mmHg)
Arm/Group | AGN-210669 Ophthalmic Solution, 0.075% | AGN-210669 Ophthalmic Solution, 0.05% | AGN-210669 Ophthalmic Solution, 0.025% | Bimatoprost Ophthalmic Solution 0.03% | AGN-210669 Vehicle Ophthalmic Solution
Number analyzed (Participants) | 35 | 33 | 33 | 30 | 36
Millimeters of Mercury (mmHg)
  Baseline - Hour 0 | 25.350 (2.8018) | 25.318 (2.9377) | 25.341 (2.6375) | 24.650 (2.0622) | 25.507 (2.9004)
  Change from Baseline at Day 14 - Hour 0 | -5.807 (3.7007) | -5.197 (3.1947) | -4.068 (2.8520) | -6.575 (3.2184) | -2.382 (2.9396)

2. Secondary Outcome: Percentage of Patients With ≥ 20% Reduction From Baseline in Diurnal IOP
Description: IOP is a measurement of the fluid pressure inside the eye. Diurnal IOP is the average of the IOP values of both eyes at each time point measured at protocol-specified times throughout the day.
Time Frame: Baseline, Day 14
Population: as for outcome 1
Measure: Number; unit: Percentage of Patients
Groups:
- AGN 210669 Non-preserved Ophthalmic Solution, 0.075%: AGN 210669 non-preserved ophthalmic solution, 0.075%. One drop in each eye each morning once-daily for 2 weeks.
Arm/Group | AGN 210669 Non-preserved Ophthalmic Solution, 0.075% | AGN-210669 Ophthalmic Solution, 0.05% | AGN-210669 Ophthalmic Solution, 0.025% | Bimatoprost Ophthalmic Solution 0.03% | AGN-210669 Vehicle Ophthalmic Solution
Number analyzed (Participants) | 35 | 33 | 33 | 30 | 36
Percentage of Patients | 62.9 | 57.6 | 30.3 | 63.3 | 2.8

ADVERSE EVENTS:
Description: The Safety Population was used to assess adverse events (AEs) and serious adverse events (SAEs), and included all patients who were randomized and received at least 1 dose of study drug.
Arm/Group | AGN-210669 Ophthalmic Solution, 0.075% | AGN-210669 Ophthalmic Solution, 0.05% | AGN-210669 Ophthalmic Solution, 0.025% | Bimatoprost Ophthalmic Solution 0.03% | AGN-210669 Vehicle Ophthalmic Solution
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/34 | 0/34 | 0/31 | 0/37
Other Adverse Events (participants affected / at risk) | 17/36 | 18/34 | 9/34 | 20/31 | 5/37
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AGN-210669 Ophthalmic Solution, 0.075% (N=36) | AGN-210669 Ophthalmic Solution, 0.05% (N=34) | AGN-210669 Ophthalmic Solution, 0.025% (N=34) | Bimatoprost Ophthalmic Solution 0.03% (N=31) | AGN-210669 Vehicle Ophthalmic Solution (N=37)
Conjunctival Hyperaemia (Eye disorders) | 10 | 11 | 5 | 12 | 3
Photophobia (Eye disorders) | 3 | 0 | 0 | 0 | 0
Eye Pain (Eye disorders) | 2 | 1 | 0 | 0 | 0
Vision Blurred (Eye disorders) | 0 | 3 | 1 | 0 | 0
Punctate Keratitis (Eye disorders) | 0 | 2 | 2 | 1 | 1
Lacrimation Increased (Eye disorders) | 1 | 0 | 1 | 2 | 1
Eye Irritation (Eye disorders) | 1 | 0 | 0 | 3 | 0
Dry Eye (Eye disorders) | 0 | 1 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.